CLINICAL TRIAL: NCT00106561
Title: A Double-Blind, Placebo-Controlled Study on the Effect of Spironolactone, in Patients With Persistent Proteinuria on Long-Term Angiotensin Converting Enzyme Inhibitor Therapy, With or With Out an Angiotensin II Receptor Blocker
Brief Title: Using the Drug Spironolactone to Test If It Reduces Protein Leakage From the Kidney
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Melbourne Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RMH2001-142
Record Dates: First submitted 2005-03-25; First posted 2005-03-28 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-03

CONDITIONS: Kidney Disease; Diabetic Nephropathy; Glomerulonephritis; Proteinuria
Keywords: spironolactone; proteinuria; angiotensin converting enzyme inhibitor; angiotensin receptor blocker; renin angiotensin aldosterone system; aldosterone
MeSH Terms: conditions — Kidney Diseases; Diabetic Nephropathies; Glomerulonephritis; Proteinuria | interventions — Spironolactone; Irbesartan

INTERVENTIONS:
Drug: Spironolactone
Drug: Irbesartan

SUMMARY:
The purpose of this study is to determine which combination of the tablets ramipril, irbesartan or spironolactone is best to lower protein leakage from the kidney.

DETAILED DESCRIPTION:
Protein leak from the kidney into the urine is an indicator of kidney damage. The higher the leak, the worse the damage and the more likely the patient will lose their kidney function long term. Interventions that lower protein leak make the kidneys last longer.

There are 2 groups of medications, both blood pressure tablets, the ACEI (angiotensin converting enzyme inhibitors) and ATRB (angiotensin receptor blockers) which have shown to reduce the amount of protein leaking from the kidney and as a result lengthen the life of the kidney. There has also been evidence that using these 2 tablets in combination is better than using either one alone. In spite of these tablets, there still remain some patients that continue to leak protein in the urine.

Recently there has been evidence that the tablet spironolactone, which is a fluid tablet, also reduces protein leakage from the kidney. In this study we look at various combinations of these tablets to see which works best to lower protein leakage from the kidney.

Patients are divided into 4 groups. Each group will receive the tablet ramipril (an ACEI). In group 1, patients will be on ramipril and 2 blank tablets, group 2 will be on ramipril, irbesartan (an ATRB) and a blank tablet, group 3 will be on ramipril, spironolactone and a blank tablet and group 4 will be on ramipril, irbesartan and spironolactone. Protein leakage is measured at the beginning and after 3 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Proteinuria more than 1.5 g/day
* On ACEI for more than 6 months
* Serum creatinine less than 200 micromol/L with less than 20% variability in the preceeding 3 months
* Creatinine clearance more than 30 ml/min, with less than 20% variability in the preceeding 3 months

Exclusion Criteria:

* Serum potassium level more than 5 mmol/L
* Treatment with corticosteroids, NSAID or immunosuppressant medication
* Acute myocardial infarction or cerebrovascular accident in the previous 6 months
* Severe uncontrolled hypertension (diastolic > 115 mmHg or systolic BP [blood pressure] > 220 mmHg)
* Evidence or suspicion of renovascular disease, obstructive uropathy, collagen disease, cancer, drug or alcohol abuse, pregnancy, or breast feeding and ineffective contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-01; Study Completion 2004-09

PRIMARY OUTCOMES:
percent reduction in 24 hour urine protein excretion

CONTACTS AND LOCATIONS:
Overall Officials: Gavin G Becker, MBBS MD, Study Director — Director Department of Nephrology, The Royal Melbourne Hospital
Locations (1):
- Department of Nephrology, The Royal Melbourne Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Chrysostomou A, Becker G. Spironolactone in addition to ACE inhibition to reduce proteinuria in patients with chronic renal disease. N Engl J Med. 2001 Sep 20;345(12):925-6. doi: 10.1056/NEJM200109203451215. No abstract available. PMID 11565535
- [Derived] Chung EY, Ruospo M, Natale P, Bolignano D, Navaneethan SD, Palmer SC, Strippoli GF. Aldosterone antagonists in addition to renin angiotensin system antagonists for preventing the progression of chronic kidney disease. Cochrane Database Syst Rev. 2020 Oct 27;10(10):CD007004. doi: 10.1002/14651858.CD007004.pub4. PMID 33107592